CLINICAL TRIAL: NCT04258865
Title: Phase I Clinical Trial to Compare the Pharmacokinetics and Tolerability of CKD-348 With Co-administration of CKD-828, D097 and D337 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Compare the Pharmacokinetics and Tolerability of CKD-348
Acronym: CKD-348
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A86_05BE1916P
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Hypertension; Dyslipidemias
Keywords: CKD-348
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: CKD-828, D097, D337 - A single oral dose of 3 tablets under fasting conditions
  Period 2: CKD-348 formulation 1 - A single oral dose of 1 tablet under fasting conditions
  Period 3: CKD-348 formulation 2 - A single oral dose of 1 tablet under fasting conditions
  Interventions: Drug: CKD-348 F1; Drug: CKD-348 F2; Drug: CKD-828, D097, D337
- Sequence 2 (Experimental): Period 1: CKD-828, D097, D337 - A single oral dose of 3 tablets under fasting conditions
  Period 2: CKD-348 formulation 2 - A single oral dose of 1 tablet under fasting conditions
  Period 3: CKD-348 formulation 1 - A single oral dose of 1 tablet under fasting conditions
  Interventions: Drug: CKD-348 F1; Drug: CKD-348 F2; Drug: CKD-828, D097, D337
- Sequence 3 (Experimental): Period 1: CKD-348 formulation 1 - A single oral dose of 1 tablet under fasting conditions
  Period 2: CKD-828, D097, D337 - A single oral dose of 3 tablets under fasting conditions
  Period 3: CKD-348 formulation 2 - A single oral dose of 1 tablet under fasting conditions
  Interventions: Drug: CKD-348 F1; Drug: CKD-348 F2; Drug: CKD-828, D097, D337
- Sequence 4 (Experimental): Period 1: CKD-348 formulation 1 - A single oral dose of 1 tablet under fasting conditions Period 2: CKD-348 formulation 2 - A single oral dose of 1 tablet under fasting conditions Period 3: CKD-828, D097, D337 - A single oral dose of 3 tablets under fasting conditions
  Interventions: Drug: CKD-348 F1; Drug: CKD-348 F2; Drug: CKD-828, D097, D337
- Sequence 5 (Experimental): Period 1: CKD-348 formulation 2 - A single oral dose of 1 tablet under fasting conditions
  Period 2: CKD-828, D097, D337 - A single oral dose of 3 tablets under fasting conditions
  Period 3: CKD-348 formulation 1 - A single oral dose of 1 tablet under fasting conditions
  Interventions: Drug: CKD-348 F1; Drug: CKD-348 F2; Drug: CKD-828, D097, D337
- Sequence 6 (Experimental): Period 1: CKD-348 formulation 2 - A single oral dose of 1 tablet under fasting conditions
  Period 2: CKD-348 formulation 1 - A single oral dose of 1 tablet under fasting conditions
  Period 3: CKD-828, D097, D337 - A single oral dose of 3 tablets under fasting conditions
  Interventions: Drug: CKD-348 F1; Drug: CKD-348 F2; Drug: CKD-828, D097, D337

INTERVENTIONS:
Drug: CKD-348 F1 — QD, PO
Drug: CKD-348 F2 — QD, PO
Drug: CKD-828, D097, D337 — QD, PO

SUMMARY:
A clinical trial to compare the pharmacokinetics and tolerability of CKD-348

DETAILED DESCRIPTION:
A randomized, open-label, single-dose, 3-way crossover clinical trial to compare the pharmacokinetics and tolerability of CKD-348 with co-administrated drugs in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19-year-old
2. Weight ≥ 50kg (man) or 45kg (woman), with calculated body mass index(BMI) of 18 to 30 kg/m2
3. Those who are eligible for adequate blood pressure criteria during screening tests Systolic blood pressure: 90 to 139 mmHg Diastolic blood pressure: 60 to 89 mmHg
4. Those who have no congenital chronic disease or chronic disease requiring treatment and who have no pathological symptoms or findings
5. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serum, urine test) and 12-lead ECG results during screening tests
6. Those who agree to contraception during the participation of clinical trial
7. Those who voluntarily decide to participate and agree to comply with the cautions after hearing and fully understanding the detailed description of this clinical trial

Exclusion Criteria:

1. Those who received investigational product or bioequivalence test drug within 6 months before the first administration of clinical trial drug
2. Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 1 month before the first administration of clinical trial drug
3. Those who donated whole blood and apheresis within 2 months or received transfusion within 1 month
4. Those who has a history of gastrointestinal surgery (
5. Those who exceeding an alcohol and smoke consumption criteria Alcohol: Men - 21 glass/week, Women - 14 glass/week (1 glass: Soju 50 mL, Beer 250mL, Wine 30mL) Smoke: 20 cigarettes/day
6. Those who has a disease history of diabetic mellitus, nephropathy, biliary obstruction, shock, dihydropyridine sensitivity, angioedema, cardiac insufficiency
7. Genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
8. Those who are deemed unfit by the investigators to participate in the clinical trial for other reasons including the results of laboratory tests
9. Women who are pregnant or who may be pregnant and breastfeed

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-348 | Pre-dose (0 hour)), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of CKD-348 | Pre-dose (0 hour)), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf of CKD-348 | Pre-dose (0 hour)), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCinf: Area under the concentration-time curve from zero up to ∞
Tmax of CKD-348 | Pre-dose (0 hour)), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Tmax: Time to maximum plasma concentration
t1/2 of CKD-348 | Pre-dose (0 hour)), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  t1/2: Terminal elimination half-life
AUCt/AUCinf of CKD-348 | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCt/AUCinf

CONTACTS AND LOCATIONS:
Overall Officials: Yook-Hwan Noh, M.D., PhD., Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea